CLINICAL TRIAL: NCT07291999
Title: Tissue Characterization in ST-Segment Elevation Myocardial Infarction: A Multicenter Registry of Patients Evaluated With Cardiac Magnetic Resonance
Brief Title: Tissue Characterization in STEMI Using Cardiac MRI: a Multicenter Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: STEMI-RMC Registry
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Ischemic Cardiovascular Disease; Magnetic Resonance
Keywords: STEMI; Cardiac magnetic resonance
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients admitted with a first STEMI treated with primary PCI, evaluated by CMR in the acute phase and follow-up

SUMMARY:
This multicenter registry includes patients with a first ST-segment elevation myocardial infarction (STEMI) who underwent cardiac magnetic resonance (CMR) imaging during the acute phase and follow-up. The registry is designed to identify clinical and CMR-derived predictors of adverse ventricular remodeling and major adverse cardiac events (MACE). CMR provides accurate and reproducible assessment of infarct size, left ventricular function, microvascular obstruction, and tissue characteristics, enabling detailed prognostic modeling.

DETAILED DESCRIPTION:
Adverse left ventricular remodeling after STEMI is a key determinant of long-term morbidity and mortality. Although primary PCI and guideline-directed therapies have improved outcomes, 10-15% of patients still develop adverse remodeling and heart failure. CMR enables precise measurement of infarct size, left ventricular volumes, ejection fraction, microvascular obstruction, and tissue parameters (T1, extracellular volume), which may enhance risk stratification compared with other imaging techniques.

The registry is based on harmonized clinical and imaging datasets from three experienced centers in Spain, forming a large repository of standardized variables. This structure facilitates the identification of predictors of infarct size, ventricular remodeling, and major adverse cardiac events (MACE), and provides a framework for the development of improved prognostic models and the exploration of potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* First STEMI evaluated within the first 24 hours of symptom onset
* At least one CMR performed during the acute phase
* Signed informed consent (for prospective patients) or previous consent (for retrospective inclusion).

Exclusion Criteria:

* Severe renal failure (GFR < 30 ml/min)
* STEMI > 24 hours after symptom onset
* Contraindications to CMR (e.g., claustrophobia, hemodynamic instability, non-MR-compatible devices, vascular clips)
* Pregnancy or breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients admitted with a first ST-segment elevation myocardial infarction (STEMI) who underwent primary percutaneous coronary intervention (PCI) and were evaluated by cardiac magnetic resonance (CMR) both in the acute phase and during follow-up. The study is conducted in tertiary academic hospitals with well-established CMR programs, ensuring standardized imaging protocols and high-quality data acquisition. Participating centers include the Hospital Clínic de Barcelona, the Hospital Clínico Universitario de Valencia, and the Hospital Universitari Vall d'Hebron, all located in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE (Major Adverse Cardiac Events) | From hospital discharge (or index CMR) to at least 6 months, with extended follow-up planned for as long as 5 years, subject to data availability.
  The primary endpoint is the occurrence of MACE during follow-up. MACE is defined as a composite of the following events:
  Cardiac death (death attributable to cardiovascular causes) Heart failure hospitalization (unplanned admission with a primary diagnosis of heart failure) Heart transplantation or durable mechanical circulatory support Appropriate ICD therapy (appropriate shock or anti-tachycardia pacing for ventricular arrhythmia in patients with implantable defibrillators).
  The occurrence of the first event in the composite will be used for time-to-event analyses.
  The first event in the composite will be used for time-to-event analyses. Event classification will be determined according to standardized definitions and based on review of available medical records.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Vall d'Hebron de Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be shared because data sharing is not planned for this study.